CLINICAL TRIAL: NCT00505609
Title: Efficacy of the Standard Days Method of Family Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SDM-IRH
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-07

CONDITIONS: Women's Health
Keywords: fertility awareness-based method; family planning; Standard Days Method; Institute for Reproductive Health; Efficacy; CycleBeads

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): The Institute for Reproductive Health trained health providers in teaching the Standard Days Method to study subjects and in study procedures. Providers counseled study participants in method use. Participants were followed for up to 13 cycles of method use.
  Interventions: Behavioral: Standard Days Method

INTERVENTIONS:
Behavioral: Standard Days Method — The Standard Days Method is a fertility awareness-based method of family planning. Users avoid unprotected intercourse during cycle days 8 to 19. Study participants were for up to 13 cycles of method use.
  Other Names: CycleBeads

SUMMARY:
The Standard Days Method® is a fertility awareness-based method of family planning in which users avoid unprotected intercourse during cycle day 8 through 19. The method is most appropriate for women with cycles that usually range 26-32 days. The clinical trial tested the contraceptive efficacy of the Standard Days Method. A total of 478 women, age 18-39 years, in Bolivia, Peru, and the Philippines, with self-reported cycles of 26-32 days, desiring to delay pregnancy at least one year were admitted to the study and followed for up to 13 cycles of method use.

DETAILED DESCRIPTION:
The Standard Days Method® is a fertility awareness-based method of family planning. Users avoid unprotected intercourse during cycle day 8 through cycle day 19. The method is most effective for women with cycles that usually range 26-32 days. It was developed by applying various formulae (i.e. various numbers of days and various sets of days) to over 7500 menstrual cycles in an existing data set from the World Health Organization, to determine which formula would provide the optimal balance between he length of the identified fertile period and the efficacy in avoiding unplanned pregnancy.

The purpose of the clinical trial was to test the efficacy of the method in preventing pregnancy.

Participants were from five sites in Bolivia, Peru, and the Philippines. In all sites, the Institute for Reproductive Health trained 5-10 health workers (service providers) in teaching the Standard Days Method to study subjects and in study procedures. Method provision involved a counseling session in which the woman (or the couple, if her partner was available) was instructed in the use of the method, and counseled on the importance of following the method recommendations to avoid pregnancy.

To assist women in monitoring their cycles, the provider gave them CycleBeads® a mnemonic device, a string of 32 beads in which each beads represents a day of the menstrual cycle. The first bead is red, representing the first day of menses; the next 6 beads are brown, representing the additional non-fertile days preceding the fertile window; the next 12 beads are white, representing days that should be considered fertile (8-19); and the remaining 13 beads are brown, again representing non-fertile days. It also has a moveable, tight-fitting rubber ring that is used to mark the current day of the cycle. Women were instructed to place the ring on the red bead on the day their menses began, and move the ring one bead per day until their menses returned. They also were told that to avoid pregnancy they should not have unprotected intercourse on the days the ring was on a white bead. If they had menstrual bleeding before day 27 of the cycle (i.e., a cycle shorter than 26 days), or if their menses had not occurred by the day after they completed all 32 beads (i.e., a cycle longer than 32 days), they were instructed to contact their provider for further assessment and advice. Women who had two cycles outside the 26 through 32 day range during the study period were advised to use another method, and were withdrawn from the study.

A total of 478 women wishing to use the Standard Days Method and meeting the eligibility criteria were admitted to the study after signing an informed consent form and interviewed monthly until they either completed 13 cycles of method use or left the study for other reasons. The first level of data collection was administered by the clients themselves. Each woman was asked to keep a daily diary to record menstrual bleeding, intercourse, and use of any other contraceptive method. The information on the diary card was reviewed by the clients and the service provider during each of the monthly follow-up contacts. In addition, follow-up forms were administered, which included questions concerning method use, satisfaction, and willingness to continue in the study.

Women who had not had their menses by day 42 of their cycle were tested for pregnancy. If results were negative, they were followed until they tested positive or their menses returned. Loss to follow-up was minimized by interviewing study participants in their homes and actively seeking out each participant, with a minimum of three attempts per cycle.

Single-decrement multi-censoring life tables were used to calculate pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18-39
* Married or living with stable partner
* At least three cycles (four periods) since last birth
* Self reported cycles 26-32 days long
* Willing to avoid intercourse 12 consecutive days every cycle
* Partners willing to collaborate
* No known infertility problems
* Not at risk for sexually transmitted infections
* No contraindications of pregnancy
* No use of hormonal contraceptives in three months prior to admission
* Desiring to avoid pregnancy for at least one year

Exclusion Criteria:

* Women who have cycles outside of the 26-32 day range
* Women/couples not interested in the method
* Women who have not yet had 3 regular cycles after childbirth
* Women who have used hormonal contraceptives in the previous 3 months
* Those women at risk for sexual transmitted infections
* Women/couples who cannot manage the fertile days by avoiding intercourse or using a barrier method

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 478 (Actual)
Dates: Start 1999-11; Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate with correct method use | 1 year (13 cycles)

SECONDARY OUTCOMES:
Pregnancy rate with typical method use | 1 year (13 cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria H. Jennings, PhD, Principal Investigator — Georgetown University
Locations (3):
- Institute for Reproductive Health, Bolivia, La Paz, Sopocachi, Bolivia
- Instituto de Salud Reporductiva, Lima, La Molina, Peru
- Institute for Reproductive Health, Philippines, Quezon City, Loyola Heights, Philippines

REFERENCES:
- [Result] Arevalo M, Jennings V, Sinai I. Efficacy of a new method of family planning: the Standard Days Method. Contraception. 2002 May;65(5):333-8. doi: 10.1016/s0010-7824(02)00288-3. PMID 12057784